CLINICAL TRIAL: NCT06698107
Title: Effectiveness of Childbirth Education Based on Salutogenic Perspective and Self-Efficacy Theory in Preventing Postpartum Depression Among Ethiopian Teenage Mothers: a Pilot RCT Study
Brief Title: Salutogenesis and Self-efficacy-based Childbirth Education Programme for Preventing Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ngai Fei Wan, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20240907003
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Depression (PPD)
Keywords: Postpartum depression; Teenage mothers; Intervention; Childbirth education
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Childbirth education programme
- Control group: (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Childbirth education programme — The intervention framework is underpinned by a converging of salutogenic and self-efficacy perspectives, aiming to enhance mothers' ability to adapt to new motherhood life despite stressors, and to address the question, "How do teenage mothers stay well despite stressful events of transition to motherhood?" The intervention consists of six sessions: three of which will be provided in the antenatal period and the other three in the postpartum period. The sessions contain two individual face-to-face educations (each lasting 60-90 minutes), two phone calls (each lasting 30 minutes), and two group discussion sessions (each lasting 90-120 minutes), as supported by the existing evidence.
  Arms: Intervention group
Other: Usual Care — The control group will receive the usual maternity care.
  Arms: Control group:

SUMMARY:
Although the transition to motherhood is often a joyful experience, there is evidence that teenage motherhood can present many stressful challenges, potentially leading to the development of postpartum depression. Postpartum depression (PPD) remains a public health issue with negative consequences for both mothers and their babies. The aim of this study is to assess the feasibility of implementing childbirth education underpinned by salutogenic and self-efficacy perspectives among teenage mothers in low-income settings. The study also aims to provide preliminary findings on the intervention's effectiveness in preventing postpartum depression among Ethiopian teenage mothers. The theoretical based childbirth education approach can enhance the psychosocial well-being of first-time teenage mothers. The intervention consists of six sessions: three during the antenatal period and three in the postpartum period. These sessions contain two individual face-to-face educations (each lasting 60-90 minutes), two phone calls (each lasting 30 minutes), and two group discussion (each lasting 90-120 minutes), as supported by the existing evidence. The study expected to support the feasibility of the study design. Preliminary findings are anticipated to show a significant difference in postpartum depression scores between the intervention and control groups, with teenage mothers in the intervention group having a lower risk of postpartum depression compared to those in the control group. Integrating sense of coherence and self-efficacy theories into maternity care services could provide empirical support for preventive efforts against postpartum depression. The findings of this study may address research gaps regarding the psychosocial wellbeing of teenage mothers, serving as baseline evidence for large scale interventional studies that consider the sociocultural and economic contexts of low-income countries.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a common mental health disorder that occur following childbirth. It typically develops within the first 12 weeks of the postpartum period, although researchers and public health experts consider PPD to be prevalent up to one year after giving birth. Although postpartum depression remains a global public health concern, it is often overlooked in the maternal healthcare system, particularly in low-and middle-income countries. The existing maternity care service often prioritizes addressing obstetrical issues while neglecting the mental well-being of labouring mothers. In Ethiopia, the prevalence of PPD among teenage mothers has reached 37%, which is much higher than the global average of 18%. Consequently, depression following childbirth continues to pose a significant risk to the overall well-being of both mothers and newborns. This study is significant in providing evidence to policymakers and health stakeholders, urging them to integrate mental health and health promotion interventions in maternity care services without imposing an additional financial burden on the healthcare system.

The role of maternity care provision during the antenatal and postnatal period is to enhance mothers' birth preparedness and complication readiness to achieve optimal maternal and infant health. However, it is crucial to practically evaluate the effectiveness of childbirth education underpinned by salutogenesis and self-efficacy perspectives in preventing PPD by enhancing mothers' sense of coherence, parenting self-efficacy, and perception of social support throughout the transition to motherhood. The findings of this study provide significant evidence for the integrating of the current disease prevention-focused approach of maternal care services with health-protective salutogenic interventions to maintain mothers' psychosocial well-being during childbirth and the parenting experience. Furthermore, the evidence may encourage countries, including Ethiopia, to implement childbirth classes that are not yet conducting in maternity care.

ELIGIBILITY:
Inclusion Criteria:

* married first-time teenage mothers aged 13-19 years attending antenatal follow-up in the selected hospitals
* a single pregnancy with 28-30 weeks of gestational age
* no pregnancy complications contraindicating vaginal delivery
* plan to have institutional delivery and postnatal visits at the selected health hospitals and who reside for a minimum of 12 weeks postdelivery around the selected hospitals

Exclusion Criteria:

* have self-reported history or current mental health problems
* participated in similar interventional programmes
* have serious medical and obstetrics problems
* having foetus with diagnosed congenital anomalies

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 6 weeks postpartum
  Edinburgh Postnatal Depression Scale is a 10-item self-report scale assessing the presence of depressive symptoms in the postnatal period. Each item is scored on a 4-point scale with total scores ranging from 0 to 30. Higher score indicates greater depressive symptoms, i.e. worse outcome.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 12 weeks postpartum
  Edinburgh Postnatal Depression Scale is a 10-item self-report scale assessing the presence of depressive symptoms in the postnatal period. Each item is scored on a 4-point scale with total scores ranging from 0 to 30. A higher score indicates greater depressive symptoms, i.e. worse outcome.
Sense of Coherence Scale | 6 weeks postpartum
  Sense of Coherence Scale is a 13-item scale assessing the extent to which teenage mothers perceive the transition to motherhood as meaningful, comprehensible and manageable. Each item is scored on a 7-point scale, with total scores ranging from 7 to 91. Higher scores indicate a stronger perception of life coherence, i.e. better outcome.
Sense of Coherence Scale | 12 weeks postpartum
  Sense of Coherence Scale is a 13-item scale assessing the extent to which teenage mothers perceive the transition to motherhood as meaningful, comprehensible and manageable. Each item is scored on a 7-point scale, with total scores ranging from 7 to 91. Higher scores indicate a stronger perception of life coherence, i.e. better outcome.
Parenting Self-Efficacy Scale | 6 weeks postpartum
  Parenting self-efficacy scale has 20 items, scored on a 4-point Likert scale, assessing teenage mothers' beliefs about their abilities to handle a set of stressful situations during the childbearing period. Higher scores indicate a stronger parenting self-efficacy, i.e. better outcome.
Parenting Self-Efficacy Scale | 12 weeks postpartum
  Parenting self-efficacy scale has 20 items, scored on a 4-point Likert scale, assessing teenage mothers' beliefs about their abilities to handle a set of stressful situations during the childbearing period. Higher scores indicate a stronger parenting self-efficacy, i.e. better outcome.
Social Support Questionnaire (modified version) | 6 weeks postpartum
  The modified version of social support questionnaire (SSQ) assessing the perceived social support during transition to motherhood, which has 6 items with 6 Likert scale points with total scores ranging from 6 to 36. Higher scores indicate a stronger perception of social support, i.e. better outcome.
Social Support Questionnaire (modified version) | 12 weeks postpartum
  The modified version of social support questionnaire (SSQ) assessing the perceived social support during transition to motherhood, which has 6 items with 6 Likert scale points with total scores ranging from 6 to 36. Higher scores indicate a stronger perception of social support, i.e. better outcome.
Perceived Stress Scale | 6 weeks postpartum
  Perceived stress scale (PSS) is a 10 items scale with 5-point Likert scoring from 0 to 4 to assess one's perceived stress level during transition to motherhood. Out of 10 items, six are negative questions (1, 2, 3, 6, 9, 10) and four are positive (4, 5, 7, 8), indicating 'perceived distress' and 'perceived coping', respectively. A higher score indicates greater perception of stress level, i.e. worse outcome.
Perceived Stress Scale | 12 weeks postpartum
  Perceived stress scale (PSS) is a 10 items scale with 5-point Likert scoring from 0 to 4 to assess one's perceived stress level during transition to motherhood. Out of 10 items, six are negative questions (1, 2, 3, 6, 9, 10) and four are positive (4, 5, 7, 8), indicating 'perceived distress' and 'perceived coping', respectively. A higher score indicates greater perception of stress level, i.e. worse outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- Ethiopia (4):
  - Addis Alem Hospital, Bahir Dar, Amhara
  - Felege Hiwot Specialized Hospital, Bahir Dar, Amhara
  - Tibebe Gion Hospital, Bahir Dar, Amhara
  - Dessie Specialized Hospital, Dessie, Amhara

IPD SHARING:
Plan to Share IPD: Undecided